CLINICAL TRIAL: NCT00904241
Title: Neuroblastoma Biology Studies
Brief Title: Biomarkers in Tumor Tissue Samples From Patients With Newly Diagnosed Neuroblastoma or Ganglioneuroblastoma
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL00B1; NCI-2009-00397 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000078642; ANBL00B1 (Other: Childrens Oncology Group); ANBL00B1 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH); UG1CA189958 (NIH); NCT00256763 (obsolete NCT alias)
Record Dates: First submitted 2009-05-16; First posted 2009-05-19 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Ganglioneuroblastoma; Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma

GROUPS / COHORTS (1):
- Ancillary-Correlative (cytology specimen collection): Patients undergo collection of blood, tissue, and bone marrow samples for analysis via RT-PCR, quantitative PCR, flow cytometry, and FISH.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in tumor tissue samples from patients with newly diagnosed neuroblastoma or ganglioneuroblastoma. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively analyze the factors that are currently used for risk-group assignment (v-myc avian myelocytomatosis viral oncogene neuroblastoma derived homolog [MYCN] copy number by fluorescent in situ hybridization [FISH], deoxyribonucleic acid [DNA] content by flow cytometry, and tumor histology using the International Neuroblastoma Pathologic Classification System) in neuroblastoma tumors at the time of diagnosis.

II. To maintain a reference bank containing clinically and genetically characterized frozen tumor tissue, tumor DNA and ribonucleic acid (RNA), histology slides and paraffin blocks, neuroblastoma-derived cell lines, patient serum and paired normal DNA obtained at the time of diagnosis, at the time of second-look surgery and at the time of relapse for future research studies.

III. To prospectively analyze 1p, 11q, 14q and 17q allelic status, MYCN copy number by quantitative polymerase chain reaction (PCR); and the expression pattern of neurotrophin-related genes in diagnostic neuroblastoma tumors, and assay for the presence of rare tumor cells in biological specimens by reverse transcription (RT)-PCR; these biological variables will be analyzed for independent clinical significance compared to MYCN amplification, International Neuroblastoma Staging System (INSS) stage, age, ploidy, and histologic variables in predicting either response to treatment or outcome.

IV. To build a database of the known biologic prognostic factors for patients on therapeutic studies.

V. To serve as a Registry for neuroblastoma patients whose tumors demonstrate clinical and genetic features defined as ?Low Risk? for treatment failure in the absence of adjuvant therapy.

SECONDARY OBJECTIVES:

I. To prospectively analyze the concordance between detection of MYCN amplification in tumor samples and quantitative detection of MYCN DNA in serum, and to analyze the prognostic significance of MYCN amplification as detected in serum samples.

II. To build a database that includes information regarding the presentation and natural history of neuroblastoma-associated health problems including but not limited to opsoclonus myoclonus ataxia (OMA) and/or spinal cord compression.

OUTLINE:

Patients undergo collection of blood, tissue, and bone marrow samples for analysis via RT-PCR, quantitative PCR, flow cytometry, and FISH.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed patients with suspected neuroblastoma, suspected ganglioneuroblastoma, or suspected ganglioneuroma/maturing subtype seen at Children's Oncology Group (COG) institutions are eligible for this study

  * There will be no penalty under any circumstances for enrollment of a patient whose definitive institutional diagnosis, or central review diagnosis, is found to be a tumor other than neuroblastoma, ganglioneuroblastoma, or ganglioneuroma/ maturing subtype
* Patients may not have received chemotherapy prior to enrollment on ANBL00B1 and procurement of study-related tissues with the following exception:

  * Patients that in the opinion of the treating physician are too ill to undergo pre-treatment tissue biopsy and require EMERGENT chemotherapy may be enrolled on ANBL00B1; documentation of the emergent nature of therapy initiation is required
* It is required that a good faith effort (documented by specimen tracking) be made to submit a neuroblastoma sample (tumor, metastasis, and/or tumor-involved bone marrow) of sufficient quality for MYCN analysis in the Neuroblastoma Reference Laboratory in order for any newly diagnosed patient to be enrolled on ANBL00B1; this should be obtained prior to initiation of therapy
* Exceptions

  * In rare cases, patients may be deemed too ill to undergo pre-treatment tissue biopsy and require EMERGENT therapy; the following eligibility guidelines apply to these cases:

    * For presumed INSS stage 4S patients: Efforts to submit tumor tissue (e.g., primary tumor, skin nodule, or metastatic site) within 96 hours of EMERGENT therapy initiation should be made; however, if the child is deemed too unstable for such a procedure they may still be enrolled as long as pre-treatment peripheral blood and serum have been submitted
    * For all other INSS stages: tumor tissue should be obtained as soon as possible within 96 hours of EMERGENT therapy initiation; patients without tumor tissues submitted within this time-frame are not eligible for enrollment

      * Note: it may not be possible to obtain all necessary tumor biomarkers for therapy stratification in such cases; if a patient enrolled on ANBL00B1 undergoes an additional diagnostic procedure within 96 hours of initiating therapy, additional tumor specimens may be submitted to obtain biomarkers used for risk classification; the decision to perform such procedures, and/or submit these specimens, is to be made by the managing clinicians and should reflect the clinical need to know the status of such biomarkers
    * Patients enrolled on ANBL1232 in Group A (either A1 or A2) will not have a tumor biopsy or resection upfront; tumor tissue submission is therefore not required for these patients to enroll on ANBL00B1; a peripheral blood and serum sample is the only specimen required to be submitted for this group of patients; should they undergo a biopsy or resection at a later date tumor can be submitted for biomarker testing at this time
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with relapsed neuroblastoma who were not enrolled on ANBL00B1 at original diagnosis are NOT eligible; samples should be submitted as part of the ABTR04B1 protocol

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2000-11-06 (Actual); Primary Completion 2100-01-01 (Estimated)

PRIMARY OUTCOMES:
Factors currently used for risk-group assignment (DNA content, MYCN copy number, and tumor histology) | Up to 3 years
  Life tables, Kaplan-Meier survival curves, log-rank tests, and Cox regression will be used to explore the relationship of laboratory variables to outcome.
Prevalence of 1p, 11q, 14q, and 17q allelic status | Up to 3 years
  These biological variables will be analyzed for independent clinical significance compared to MYCN amplification, INSS stage, age, ploidy, and histologic variables in predicting either response to treatment or outcome.
MYCN copy number by quantitative PCR | Up to 3 years
  These biological variables will be analyzed for independent clinical significance compared to MYCN amplification, INSS stage, age, ploidy, and histologic variables in predicting either response to treatment or outcome.
Expression pattern of neurotrophin-related genes in diagnostic neuroblastoma tumors | Up to 3 years
  These biological variables will be analyzed for independent clinical significance compared to MYCN amplification, INSS stage, age, ploidy, and histologic variables in predicting either response to treatment or outcome.
Presence of rare tumor cells in biological specimens by RT-PCR | Up to 3 years
  These biological variables will be analyzed for independent clinical significance compared to MYCN amplification, INSS stage, age, ploidy, and histologic variables in predicting either response to treatment or outcome.
Database of the known biologic prognostic factors for patients on therapeutic studies | Up to 3 years
  During the testing for treatment effect in Phase III trials, the biologic prognostic factors may be needed for adjustment in the Cox regression model-building process.

SECONDARY OUTCOMES:
MYCN status per tumor | Up to 3 years
  Cross tabulations of MYCN status per tumor versus MYCN status per blood will be generated, the percentage concordant and the percentage discordant will be calculated, and receiver operating characteristic (ROC) analyses will be performed. Kaplan-Meier curves of MYCN status per blood will be generated, and a logrank test comparison performed. The prognostic ability of MYCN status per tumor versus MYCN status per blood will be tested in a multivariable Cox model.
MYCN status per blood | Up to 3 years
  Cross tabulations of MYCN status per tumor versus MYCN status per blood will be generated, the percentage concordant and the percentage discordant will be calculated, and ROC analyses will be performed. Kaplan-Meier curves of MYCN status per blood will be generated, and a logrank test comparison performed. The prognostic ability of MYCN status per tumor versus MYCN status per blood will be tested in a multivariable Cox model.
Incidence of OMA | Up to 3 years
  Descriptive analysis will be performed.
Incidence of spinal cord compression | Up to 3 years
  Descriptive analysis will be performed.
Presentation with multifocal primary tumors | Up to 3 years
  Descriptive analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hogarty, Principal Investigator — Children's Oncology Group
Locations (259):
- United States (223):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cardon Children's Medical Center, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (10):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- University Medical Center Groningen, Groningen, Netherlands
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- Switzerland (3):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Derived] Furner B, Cheng A, Desai AV, Benedetti DJ, Friedman DL, Wyatt KD, Watkins M, Volchenboum SL, Cohn SL. Extracting Electronic Health Record Neuroblastoma Treatment Data With High Fidelity Using the REDCap Clinical Data Interoperability Services Module. JCO Clin Cancer Inform. 2024 May;8:e2400009. doi: 10.1200/CCI.24.00009. PMID 38815188